CLINICAL TRIAL: NCT05055336
Title: Longitudinal Evaluation of Gastric Emptying and Accommodation in Children With Dyspepsia: Toward Individualized Care in Functional Abdominal Pain Disorders
Brief Title: Longitudinal Evaluation of Gastric Emptying and Accommodation in Children With Dyspepsia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution.
Sponsor: University of Miami (Other)
Collaborators: American Neurogastroenterology and Motility Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20210662
Record Dates: First submitted 2021-08-23; First posted 2021-09-24 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Gastroparesis; Dyspepsia
MeSH Terms: conditions — Gastroparesis; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastroparesis (Experimental): Participants in this group are children diagnosed with gastroparesis per gastric emptying scintigraphy. Participants will be receiving a gastric emptying breath test three times over the course of 6 months and an ultrasound of the stomach once.
  Interventions: Other: Gastric emptying breath test; Other: Stomach ultrasound
- Dyspepsia (Experimental): Participants in this group are children diagnosed with functional dyspepsia per gastric emptying scintigraphy. Participants will be receiving a gastric emptying breath test three times over the course of 6 months and an ultrasound of the stomach once.
  Interventions: Other: Gastric emptying breath test; Other: Stomach ultrasound
- Healthy Controls (Experimental): Participants in this group are children that do not have gastroparesis, functional dyspepsia, or any other gastroenterology condition. Participants will be getting an ultrasound once.
  Interventions: Other: Stomach ultrasound

INTERVENTIONS:
Other: Gastric emptying breath test — The gastric emptying breath test is used to diagnose gastroparesis. Participants ingest spirulina in a meal and samples are taken every 45 minutes for 4 hours.
  Arms: Dyspepsia; Gastroparesis
Other: Stomach ultrasound — Ultrasound of the fundus of the stomach will be done immediately after ingestion of the test meal, at 15 minutes, and at 30 minutes.

SUMMARY:
The purpose of this research is to further study the relationship between gastroparesis (GP) (a condition in which the stomach cannot empty itself of food in a normal fashion) and functional dyspepsia (FD) (frequent symptoms of indigestion that have no obvious cause).

ELIGIBILITY:
Inclusion Criteria:

* Able to complete the Pediatric Cardinal Symptoms Questionnaire
* Both parent and child must be able to speak and understand English or Spanish

Exclusion Criteria:

* Have global developmental delay, autism disorder, or psychosis
* Are nonverbal and/or illiterate
* Lack fluency in English or Spanish
* Have other GI comorbidities such as inflammatory bowel disease, celiac disease, eosinophilic esophagitis, peptic ulcer disease, GI malignancy, or gastroesophageal reflux disease responsive to medications (medical records will be reviewed to detect these exclusions)
* Have a history of surgical procedures that could have potentially affected their GI tract anatomy, such as fundoplication or Ladd's procedure.
* Healthy child presenting to their well child care visit must not report a history of dyspepsia, have a history of any gastrointestinal disease, or be taking any medication that can disturb the GI tract motility.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying rate | up to 6 months
  As measured by the spirulina breath test

SECONDARY OUTCOMES:
Percentage of food retained in the stomach | Day 1
  Fundic accommodation will be reported as the percentage of food retained in the fundus using an ultrasound before and after meal ingestion.
Pediatric Cardinal Symptoms Questionnaire Scores | Up to 6 months
  The pediatric symptoms questionnaires has a total score ranging from 0-600. Higher score means worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Liz Febo-Rodriguez, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No